CLINICAL TRIAL: NCT01191138
Title: Randomized Control Trial Comparing Gastric Emptying Following Infracolic vs Supracolic Gastrojejunostomy After Whipples Pancreaticoduodenectomy
Brief Title: Gastric Emptying After Infracolic or Supracolic Gastrojejunostomy Following Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: KK Nuclear Scan (Unknown)
Responsible Party: Pradeep Rebala, Asian Institute of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AIG-GIS-20090
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Postprocedural Gastric Stasis
Keywords: Delayed Gastric emptying; Gastric emptying scintigraphy; Pancreatic fistula; Pancreatic Neoplasms; Whipple Operation
MeSH Terms: conditions — Gastroparesis; Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infracolic Anastamosis (Other): The gastrojejunal anastamosis is done in the infracolic compartment
  Interventions: Procedure: Infracolic gastrojejunal anastamosis
- Supracolic Anastamosis (Other): The gastrojejunal anastamosis is done in the supracolic compartment
  Interventions: Procedure: Supracolic gastrojejunal anastamosis

INTERVENTIONS:
Procedure: Infracolic gastrojejunal anastamosis — Following resection in whipples pancreaticoduodenectomy, the gastrojejunal anastamosis is done in the infracolic compartment by bringing down the stomach below the mesocolon to the left of the middle colic artery
  Other Names: Infracolic and retrocolic Gastrojejunostomy
  Arms: Infracolic Anastamosis
Procedure: Supracolic gastrojejunal anastamosis — Following resection in whipples pancreaticoduodenectomy, the gastrojejunal anastamosis is done in the supracolic compartment.
  Other Names: Supracolic and retrocolic gastrojejunostomy
  Arms: Supracolic Anastamosis

SUMMARY:
Patients undergoing whipples pancreaticoduodenectomy tend to develop delayed gastric emptying.

The study compares two types of anastamosis of stomach to jejunum (supracolic and infracolic) and compares whether it influences the gastric emptying.

The clinical evidence of delayed gastric emptying is correlated with objective evidence of liquid and solid emptying by radionuclide study.

The study also tries to evaluate whether pancreatic leak correlates with delayed gastric emptying

DETAILED DESCRIPTION:
METHODOLOGY:

This randomized control trial includes all patients undergoing whipples pancreaticoduodenectomy st Asian Institute of Gastroenterology. All patients were randomized by a closed envelope technique. The envelope was opened after complete resection of the specimen and then allocating the patients into either of the two groups, Group A- Infracolic Gastrojejunostomy, Group B- Supracolic Gastrojejunostomy.

Inclusion Criteria:

* All patients undergoing whipples pancreaticoduodenectomy, who consented for the trial and found to be resectable at surgery.

Exclusion Criteria:

* Unresectable tumors at surgery
* Patients in whom gastric emptying studies could not be done due to any reason
* Documented Mechanical obstruction at Gastrojejunal anastamosis
* Post operative mortality due to other causes

After the resection, a Roux loop of jejunum is prepared and taken up through a rent in the transverse mesocolon to which an end to side Hepaticojejunostomy followed by Pancreaticojejunostomy is done in both the groups.

In Group A Infracolic gastrojejunostomy is done in the infracolic compartment to the same loop of jejunum after pulling the stomach down through another rent in the transverse mesocolon to the left of middle colic artery, thereby compartmentalizing or separating gastrojejunostomy from Hepaticojejunostomy and pancreaticojejunostomy.

In Group B Supracolic gastrojejunostomy is done in the supracolic compartment to the same Roux loop of jejunum.

All the patients undergo a feeding jejunostomy. Postoperatively all the patients were managed according to a standard protocol, daily monitoring of Ryle's tube output and drain fluid output was recorded. Drain fluid amylase levels and serum amylase levels were estimated on postoperative day 3, 5 and 7. Ryle's tube was removed if the output was <200ml in 24hrs after confirming that the tube was patent.

Oral feeds were started after removal of Ryle's tube, initially with liquids followed by semisolids and then normal diet. Patient's daily intake is recorded. Any adverse event of vomiting, abdominal distension and succussion splash was recorded by the person blinded about the technique of anastamosis. If there was clinical suspicion of gastric outlet obstruction, Ryle's tube was placed and output recorded. If mechanical cause for gastric outlet obstruction was suspected, then contrast study and/or gastroscopy was done to confirm.

Graded enteral nutrition was started in all the patients from post operative day 3 through the feeding jejunostomy tube.

Any medications effecting GI motility were avoided till the gastric emptying studies were performed

Clinically delayed gastric emptying was defined according to International study group of pancreatic Surgeons (ISGPS), as Grade A, B and C. Pancreatic fistula was defined based on International Study Group on Pancreatic Fistula (ISGPF) as Grade A, B and C.

Radio isotope gastric emptying studies were done for both liquids and solids on postoperative day 7 & 8 respectively. Test was performed and interpreted by the investigator who is blinded about the type of anastamosis.

At the end the groups will be analyzed whether they were comparable with regard to the age, sex and diagnosis. The gastric emptying (Clinical, liquid meal and solid meal emptying) will be compared between both procedure groups. Correlation of clinical evidence of gastric emptying with liquid and solid emptying is calculated. Correlation of pancreatic anastomotic leak with gastric emptying is also done.

PROTOCOL OF GASTRIC EMRTYING STUDY:

Liquid study on one day & solid study on the next day

Tracer to be use:

1. Tc99m-DTPA in water 400ml for 70 Kg adult; volume to be adjusted based on patient weight, is used for liquid emptying study.
2. Tc99m-Pertechnetate labeled with Idly during cooking, 300gm for 70 Kg adult; volume to be adjusted based on patient weight, is used for solid emptying study.

IMAGING TECHNIQUE:

Sequential static images are to be obtained with patient in erect position from anterior & posterior projections of the abdomen Liquids - 1min image for every 15min for 90mins (to be extended to 120 mins if necessary).

Solids - 1min image for every 30min for 4hrs (to be extended if necessary).

IMAGE PROCESSING:

Region of interest to be generated over stomach region, after verifying with the surgeon initially for standardization Now Geometric mean of counts calculated from the stomach and used to generate the time activity curve, percentage emptying at different time intervals and T1/2 to be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Whipples procedure

Exclusion Criteria:

* Unresectable tumors at surgery
* Postoperative mechanical obstruction
* Postoperative mortality, where the test could not be done

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying assessed clinically and correlated objectively with liquid and solid emptying of radionucleotide | 30 days after surgery
  Gastric emptying in the postoperative period in the form of tolerence of food and removal of ryles tube is assessed. This is correlated with liquid and solid emptying of radionucleotide

SECONDARY OUTCOMES:
Correlation of pancreatic duct leak with gastric emptying | 30 days after surgery
  The pancreatic duct leak is correlated with gastric emptying

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Rebala, MS., M Ch, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute Of Gastroenterology India, Hyderabad, Andhra Pradesh, India